CLINICAL TRIAL: NCT05421910
Title: Clinical Feasibility of ROBERT-SAS in Severely Impaired Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roessingh Research and Development (Other)
Collaborators: Aalborg University (Other); Lifescience-Robotics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: NL80574.000.22
Record Dates: First submitted 2022-06-09; First posted 2022-06-16 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Stroke
Keywords: Robotic; Electrical stimulation; Lower extremity; Stroke
MeSH Terms: conditions — Stroke | interventions — Electric Stimulation

STUDY DESIGN:
Intervention Model Description: One group will receive robotic training as soon as possible, another group will receive robotic training 3-5 weeks, after submission to the rehab center. Normal rehabilitation will also carry on.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early training group (Experimental): The early group will receive robotic training combined with electrical stimulation as soon as possible after submission to the rehab center. With a frequency of three times a week for 3-5 weeks, dependent on the capabilities of the patients.
  Interventions: Device: robotic training combined with electrical stimulation
- Late training group (Active Comparator): The late training group will receive robotic training combined with electrical stimulation 3-5 weeks after submission to the rehab center. With a frequency of three times a week for 3-5 weeks, dependent on the capabilities of the patients.
  Interventions: Device: robotic training combined with electrical stimulation

INTERVENTIONS:
Device: robotic training combined with electrical stimulation — Active training of movements in supine position. Movements such as knee extension and ankle dorsal flexion.

SUMMARY:
Robotic training can be used to provide intensive training during the (early phases of) rehabilitation of a stroke. ROBERT®-SAS training is designed to create an active and intensive training tool for the rehabilitation of the lower extremity of stroke patients. Currently this has only be tested in a lab-based setting, which showed that is was feasible and could be executed while still being comfortable for the patient. The next step will be implementing the device in a clinical setting. Therefore, aims the current study to assess the feasibility of ROBERT®-SAS training in clinical setting, in acute stroke patients.

DETAILED DESCRIPTION:
Rationale: Stroke is one of the leading causes of disability of adults in the European Union. Around 80% of stroke survivors experience deficits in motor control, resulting in problems with keeping balance and walking, for instance. The extent and amount of deficits differ per individual. Interventions to train the lower extremity almost always consist of walking exercises. However, patients in the acute phase or with severely affected lower extremity function are often unable to walk or to walk independently. Therefore, the combination of a robot (ROBERT®) and functional electrical stimulation (ES) is being developed to provide a training tool for early rehabilitation. In the current study a combination of robot and ES will be evaluated in clinical setting.

Objective: The primary objective of the current study is to assess the feasibility of ROBERT®-SAS training in clinical setting, in acute stroke patients, including patient and therapist perspectives.

Study design: The current study is an observational study.

Study population: In the current study ten (sub) acute stroke patient will be included, with severely affected lower extremity. Five of these ten will be included as soon as possible after arrival at the rehabilitation centre. Another five will be included 3-5 weeks after arrival/start of the rehabilitation.

Main study parameters/endpoints: The main outcome parameter is the SUS score from both the patients and the therapists.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The current study consists of several measurement sessions in Roessingh Rehabilitation Centre, during the normal rehabilitation time. The robot, ROBERT® is CE-certified. However, the combination ROBERT®-SAS, combining both ES and robot support, is not, although previous tests have shown this approach is possible and tolerable by healthy persons and stroke patients. The risks are regarded as minimal because it is without invasive procedures, with room for rest in between trial sets as required by the participant, and application of individual stimulation profiles to not exceed tolerance levels or inflict pain during electrostimulation.

ELIGIBILITY:
Inclusion Criteria:

* Sub(acute) stroke (< 6 months post-stroke)
* Above 18 years
* Able to provide informed consent
* An ischemic or haemorrhagic stroke
* Hemiparetic lower extremity

Exclusion Criteria:

* Premorbid disability of lower extremity
* Severe cognitive impairment, unable to follow simple instructions and unable to understand Dutch.
* Skin lesions at the hemiparetic leg
* Progressive neurological diseases (i.e. Parkinson, dementia, etc.)
* Contraindication for mobilization like unhealed lower limb fracture
* Use of pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
System Usability Scale (SUS) score | 15 minutes
  The System Usability Scale of patients and therapists. 10 questions with a 5-point response scale. The total score can range from 0 - 100, in which a higher score indicates a better usability

SECONDARY OUTCOMES:
Electromyography (EMG) | 30 minutes
  Surface EMG of the muscle that will be stimulated with electrical stimulation, expressed in volt.
Force | 30 minutes
  Resulting force measured with the robot, expressed in kg
Frequency | 30 minutes
  As a settings of the stimulation expressed in Hertz
Assist-As-Needed (AAN) stages | 30 minutes
  The trajectory completion rate for the different stages of AAN. (different types of assistance). There are three different types, no assistance, electrical stimulation assistance and an combination of electrical stimulation and robot support.
Fugl-Meyer Assessment (FMA) | 10 minutes
  Lower extremity module, to assess leg function. Scores can range between 0 and 28, in which a higher score indicates a higher leg function.
Motricity Index (MI) | 10 minutes
  Lower extremity part, to assess the leg function. Scored for Ankle, knee and hip separately between 0 - 33 in which zero is know movement and 33 is normal movement. Total score can range between 0 - 99. (summation of the three joints)
Functional Ambulation Categories (FAC) | 5 minutes
  To assess the walking capabilities, score between 0 and 5, in which 5 indicates a better walking capability.
Type of movement | 30 minutes
  Type of movement that will be trained during the measurements. Can be knee extension or ankle dorsal flexion with electrical stimulation.
Questionnaire Experience | 15 minutes
  Questions about their experience with ROBERT for all stakeholders. Open questions which will not have a score, but will be interpreted on question level.
Pulse width of the electrical stimulation | 30 minutes
  As a settings of the stimulation expressed in milliseconds
Amplitude of the electrical stimulation | 30 Minutes
  As a settings of the stimulation expressed in milliampere
Amount of repetitions | 30 minutes
  The amount of repetitions during one set of a specific movement.
Resistance level | 30 minutes
  The amount of resistance during the training, can be changed during a set if necessary. The resistance can differ between 0-10, in which 10 is the heaviest.

OTHER OUTCOMES:
Gender | 1 minutes
  gender will be noted as subject characteristic
Age | 1 minutes
  Age will be noted as subject characteristic in years
Time since stroke | 1 minutes
  time science stroke will be noted as subject characteristic in months
Weight | 1 minutes
  Weight will be noted as subject characteristic and used for BMI calculation, noted in kg
Height | 1 minutes
  Height will be noted as subject characteristic and used for BMI calculation, noted in meters
Affected side | 1 minutes
  The affected side will be used as subject characteristic

CONTACTS AND LOCATIONS:
Overall Officials: Gerdienke Prange, PhD, Principal Investigator — Roessingh Research and Development
Locations (1):
- Roessingh Research and Development, Enschede, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No